CLINICAL TRIAL: NCT02955329
Title: Vaping THC From Electronic Cigarettes: a Novel Evaluation of Intake and Pharmacokinetics
Brief Title: Vaping THC From Electronic Cigarettes
Acronym: V-PAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 18-24854; 3R01DA039264-02S1 (NIH)
Record Dates: First submitted 2016-10-31; First posted 2016-11-04 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Marijuana Dependence
Keywords: THC; Tobacco; Vaping
MeSH Terms: conditions — Marijuana Abuse; Vaping | interventions — Nicotine; Tobacco Products; nabiximols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Tobacco Arm (Experimental): Participants will vape tobacco leaves with nicotine out of the PAX device.
  Interventions: Drug: Nicotine; Device: PAX Loose Leaf Vaporizer
- Cannabis Arm (Experimental): Participants will vape marijuana leaves with THC (Tetrahydrocannabinol) out of the PAX device.
  Interventions: Drug: Cannabis; Device: PAX Loose Leaf Vaporizer
- Combined Cannabis and Tobacco Arm (Experimental): Participants will vape flavorless 6% nicotine e-liquid, followed by THC (Tetrahydrocannabinol) out of the PAX device.
  Interventions: Drug: Nicotine; Drug: Cannabis; Device: PAX Loose Leaf Vaporizer

INTERVENTIONS:
Drug: Nicotine — Participants will vape tobacco leaves with nicotine out of the PAX device.
  Other Names: Tobacco Leaf
  Arms: Combined Cannabis and Tobacco Arm; Tobacco Arm
Drug: Cannabis — Participants will vape marijuana leaves with nicotine out of the PAX device.
  Other Names: Marijuana Leaf
  Arms: Cannabis Arm; Combined Cannabis and Tobacco Arm
Device: PAX Loose Leaf Vaporizer — In all three arms, the participant will be using the same PAX electronic cigarette device. The only difference is whether the participant will be vaping nicotine only, THC only, or nicotine and THC.

SUMMARY:
This study aims to understand THC pharmacology and the safety of cannabis vaping, including the pharmacology and safety of co-administration of nicotine and THC. The study is designed as a within-subjects single-blinded crossover study. Fourteen smokers of tobacco cigarettes and cannabis will switch between three conditions, namely: (a) vaping cannabis leaf, (b) vaping tobacco containing nicotine and (c) vaping a combination of cannabis leaf and tobacco containing nicotine. All participants will vape each product with the PAX loose-leaf vaporizer. The study will be conducted during three outpatient visits separated by at least 48 hours. The order of treatment (cannabis leaf, tobacco with nicotine, cannabis leaf & tobacco with nicotine) will be counterbalanced between subjects. Subjects will be blinded to the content of the vaporizer on the study day but will be told during screening that they will vape cannabis alone, tobacco alone, and cannabis plus tobacco with nicotine.

DETAILED DESCRIPTION:
Electronic cigarettes (e-cigarettes) have proliferated at a rapid rate since their introduction into the US market in 2007, and their use as a form of nicotine delivery far outpaced the science base. Although the design of these devices continues to evolve, we have previously described nicotine intake, systemic retention, pharmacokinetics, and vaping behavior associated with self-administration of e-cigarettes. We demonstrated that while the shape of the plasma nicotine concentration-time curve for e-cigarettes is similar to tobacco cigarettes, the maximum plasma nicotine concentration is, on average, lower for e-cigarettes. During ad libitum access, e-cigarettes were vaped intermittently in groups of 2-5 puffs or single puffs such that plasma nicotine levels rose gradually and peaked at the end of the 90-minute session. This differs from the rapid increase in plasma nicotine observed during controlled use of e-cigarettes or during tobacco cigarette smoking. Taken together, these results indicate that e-cigarettes have the potential to produce and sustain nicotine addiction but their use and abuse liability may differ from tobacco cigarettes.

The study is designed as a within-subjects, single-blinded crossover study. Fourteen smokers of tobacco cigarettes and cannabis will switch between three conditions, namely: (a) vaping cannabis leaf, (b) vaping tobacco containing nicotine and (c) vaping a combination of cannabis leaf and tobacco containing nicotine. All participants will vape each product with the PAX loose-leaf vaporizer, which will be purchased by the study team. The cannabis leaf will be obtained through the National Institute on Drug Abuse Drug Supply Program. The tobacco-containing nicotine, used in conditions (b) and (c) will come from commercially available Marlboro brand cigarettes. The same amount of cannabis or tobacco will be used in all conditions.

The study will be conducted during three outpatient visits separated by at least 48 hours. The order of treatment (cannabis leaf, tobacco with nicotine, cannabis leaf & tobacco with nicotine) will be counterbalanced between subjects. Subjects will be blinded to the content of the vaporizer on the study day but will be told during screening that they will vape cannabis alone, tobacco alone, and cannabis plus tobacco with nicotine.

While scientists struggle to keep up with the latest electronic cigarette trends, the use of these devices for cannabis rather than nicotine is increasingly prevalent. Electronic cigarette use is not restricted to nicotine. Marijuana, the most widely used illicit drug has traditionally been combusted but the vaping of loose-leaf marijuana and THC oil has been increasing. the latest national data show that 7.6% of current marijuana users (past 30 days) and 9.9% of ever cannabis users (lifetime) administered THC through a vaporizer or electronic device (the study did not differentiate between vaporizers and electronic devices like e-cigarettes). The prevalence of vaped marijuana or THC is higher among younger adults. Prevalence of vaped marijuana/THC among 18-24 and 25-34 year-old ever marijuana users was 19.3% and 16.3%, respectively, compared to 8.8% for 35-49 year-olds and 5.7% for those 50 years and over. A recent study also showed high rates of cannabis vaping among high school students (18.0% among ever e-cigarette users). Smoking of a combination of tobacco and marijuana in cigarette form is also common, particularly in Europe. However, very little is known about the safety and pharmacokinetics of this co-administration making it a critical area of research.

ELIGIBILITY:
Inclusion

* Age >=21 years <=70 years
* Regular user of tobacco cigarettes (daily or most days)
* Regular user of cannabis in any form (combusted or ingested) at least 5 days out of the month.
* Positive for Tetrahydrocannabinol (THC) on screening toxicology test
* Willing to abstain from tobacco smoking and all other combustible products (ex: cigars) for 12 hours prior to each outpatient hospital admission.
* Willing to abstain from smoking/ingesting cannabis for 12 hours prior to each outpatient hospital admission.
* Willing to abstain from using any kind of nicotine products for 12 hours prior to each outpatient hospital admission (ex: electronic cigarettes, nicotine replacement therapy).
* Saliva cotinine ≥ 30 ng/mL and/or NicAlert of 6
* Healthy (based on limited physical examination and medical history collected during screening)
* Heart rate < 105 beats per minute (BPM)
* Systolic Blood Pressure < 160 and > 90 (considered out of range if both machine and manual readings are above/below these thresholds)
* Diastolic Blood Pressure < 100 and > 50 (considered out of range if both machine and manual readings are above/below these thresholds)
* Body Mass Index ≤<=38.0

Exclusion

* Medical (The following unstable medical conditions):
* Heart disease
* Uncontrolled hypertension
* Thyroid disease (okay if controlled with medication)
* Diabetes
* Hepatitis B or C or Liver disease
* Glaucoma
* Prostatic hypertrophy
* History of paranoia after marijuana use
* Psychiatric conditions
* Current or past schizophrenia, and/or current or past bipolar disorder
* Adult onset Attention-deficit/hyperactivity disorder (ADHD) (if being treated)
* Participants with current or past depression and/or anxiety disorders will be reviewed by the study physician and considered for inclusion
* History of psychiatric hospitalizations are not exclusionary, but study participation will be determined as per study physician's approval
* Drug/Alcohol Dependence
* Alcohol or illicit drug dependence within the past 12 months with the exception of those who have recently completed an alcohol/drug treatment program and are currently abstaining from drug and alcohol
* Positive toxicology test at the screening visit (THC & prescribed medications okay)
* Methadone replacement therapy
* Scoring a 2 or higher on the Severity of Dependence Scale for cannabis use.
* Psychiatric medications
* Current regular use of any psychiatric medications with the exception of Selective Serotonin Reuptake Inhibitors (SSRIs) and serotonin-norepinephrine reuptake Inhibitors (SNRIs) and current evaluation by the study physician that the participant is otherwise healthy, stable, and able to participate.
* Other Medications
* Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, dexamethasone, phenobarbital, and other anticonvulsant drugs).
* Concurrent use of nicotine-containing medications
* Other/Misc. Chronic Health Conditions
* Oral thrush
* Fainting
* Untreated thyroid disease
* Other "life threatening illnesses" as per study physician's discretion
* Use of Other Tobacco Products (OTP); any of the following products in combination more than 15 times in the past month
* smokeless tobacco
* pipes
* cigars, cigarillos
* blunts, spliffs
* Pregnancy
* Pregnancy (self-reported and urine pregnancy test)
* Breastfeeding (determined by self-report)
* Concurrent participation in another clinical trial
* Inability to communicate in English
* Planning to quit smoking or cannabis use within the next 60 days

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King BA, Patel R, Nguyen KH, Dube SR. Trends in awareness and use of electronic cigarettes among US adults, 2010-2013. Nicotine Tob Res. 2015 Feb;17(2):219-27. doi: 10.1093/ntr/ntu191. Epub 2014 Sep 19. PMID 25239961
- [Background] Arrazola RA, Singh T, Corey CG, Husten CG, Neff LJ, Apelberg BJ, Bunnell RE, Choiniere CJ, King BA, Cox S, McAfee T, Caraballo RS; Centers for Disease Control and Prevention (CDC). Tobacco use among middle and high school students - United States, 2011-2014. MMWR Morb Mortal Wkly Rep. 2015 Apr 17;64(14):381-5. PMID 25879896
- [Background] St Helen G, Havel C, Dempsey DA, Jacob P 3rd, Benowitz NL. Nicotine delivery, retention and pharmacokinetics from various electronic cigarettes. Addiction. 2016 Mar;111(3):535-44. doi: 10.1111/add.13183. Epub 2015 Nov 11. PMID 26430813
- [Background] St Helen G, Ross KC, Dempsey DA, Havel CM, Jacob P 3rd, Benowitz NL. Nicotine Delivery and Vaping Behavior During ad Libitum E-cigarette Access. Tob Regul Sci. 2016 Oct;2(4):363-376. doi: 10.18001/TRS.2.4.8. PMID 28393086
- [Background] Center for Behavioral Health Statistics and Quality. Behavioral health trends in the United States: Results from the 2014 National Survey on Drug Use and Health. NSDUH; 2015.
- [Background] Schauer GL, King BA, Bunnell RE, Promoff G, McAfee TA. Toking, Vaping, and Eating for Health or Fun: Marijuana Use Patterns in Adults, U.S., 2014. Am J Prev Med. 2016 Jan;50(1):1-8. doi: 10.1016/j.amepre.2015.05.027. Epub 2015 Aug 12. PMID 26277652
- [Background] Morean ME, Kong G, Camenga DR, Cavallo DA, Krishnan-Sarin S. High School Students' Use of Electronic Cigarettes to Vaporize Cannabis. Pediatrics. 2015 Oct;136(4):611-6. doi: 10.1542/peds.2015-1727. Epub 2015 Sep 7. PMID 26347431
- [Background] Akre C, Michaud PA, Berchtold A, Suris JC. Cannabis and tobacco use: where are the boundaries? A qualitative study on cannabis consumption modes among adolescents. Health Educ Res. 2010 Feb;25(1):74-82. doi: 10.1093/her/cyp027. Epub 2009 Jun 10. PMID 19515745
- [Background] Amos A, Wiltshire S, Bostock Y, Haw S, McNeill A. 'You can't go without a fag...you need it for your hash'--a qualitative exploration of smoking, cannabis and young people. Addiction. 2004 Jan;99(1):77-81. doi: 10.1111/j.1360-0443.2004.00531.x. PMID 14678065

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 8 total participants received all 3 interventions over the course of 3 days, with the sequence of the interventions varied for each participant. The order of treatment (cannabis leaf, tobacco with nicotine, cannabis leaf & tobacco with nicotine) will be counterbalanced between subjects
Groups:
- All Participants: All participants were enrolled and received each of the interventions in a different order. Each intervention lasted 1 day.
Period: Tobacco Arm
Arm/Group | All Participants
Started (Participants vaped tobacco leaves with nicotine out of the PAX device.) | 8
Completed | 8
Not Completed | 0
Period: Cannabis Arm
Arm/Group | All Participants
Started (Participants vaped marijuana leaves with Tetrahydrocannabinol (THC) out of the PAX device) | 8
Completed | 8
Not Completed | 0
Period: Combined Cannabis and Tobacco Arm
Arm/Group | All Participants
Started (Participants vaped flavorless 6% nicotine e-liquid, followed by THC out of the PAX device.) | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Delivered and Retained Doses
Description: Delivered Tetrahydrocannabinol (THC) and nicotine doses are estimated as the change in e-cigarette weight × concentration of THC or nicotine in e-liquid. The amount of THC or nicotine systemically retained is estimated as delivered dose minus amount in gas traps.
Time Frame: Study Day 1-3
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
grams (g) | 0.016 (0.003) | 0.018 (0.008) | 0.026 (0.008)

2. Primary Outcome: Median Peak THC Concentration (Cmax)
Description: Median peak concentration of THC between vaped loose-leaf cannabis, mixture of cannabis and tobacco containing nicotine, and the tobacco alone treatment condition will be reported
Time Frame: Study Day 1-3
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
mg/mL | 1.52 [0.90 to 2.14] | 9.72 [7.43 to 12.01] | 25.74 [20.8 to 30.68]

3. Primary Outcome: Median Peak Nicotine Concentration (Cmax)
Description: Median peak concentration of nicotine between vaped loose-leaf cannabis, mixture of cannabis and tobacco containing nicotine, and the tobacco alone treatment condition will be reported
Time Frame: Study Day 1-3
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 0.55 [0.43 to 0.67] | 0.38 [0.10 to 0.66] | 1.59 [1.34 to 1.84]

4. Primary Outcome: Median THC Exposure
Description: Median exposure of nicotine using area under the blood/plasma concentration-time curve(AUC) between vaped loose-leaf cannabis, mixture of cannabis and tobacco containing nicotine, and the tobacco alone treatment condition will be reported
Time Frame: Study Day 1-3
Measure: Median (Inter-Quartile Range); unit: ng/mL•minute
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
ng/mL•minute | 201.6 [108.4 to 294.8] | 306.4 [215.4 to 397.5] | 585.6 [388.2 to 783.0]

5. Primary Outcome: Median Nicotine Exposure
Description: Compare median exposure of nicotine using AUC (area under the blood/plasma concentration-time curve) between vaped loose-leaf tobacco containing nicotine vs. mixture of cannabis and tobacco containing nicotine.
Time Frame: Study Day 1-3
Measure: Median (Inter-Quartile Range); unit: ng/mL•minute
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
ng/mL•minute | 63.1 [54.1 to 72.1] | 42.7 [7.4 to 78.0] | 134.9 [122.2 to 147.5]

6. Primary Outcome: Mean Heart Rate
Description: Heart rate monitoring by pulse oximeter
Time Frame: Study Day 1-3
Measure: Mean (95% Confidence Interval); unit: bpm
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
bpm | 67.3 [65.5 to 69.1] | 66.8 [64.5 to 69.1] | 70.5 [68.4 to 72.6]

7. Primary Outcome: Mean Score on the Drug Effects Questionnaire (DEQ)
Description: The Drug Effects Questionnaire (DEQ) is widely used in studies of acute subjective response (SR) to a variety of substances which assessed the extent to which participants (1) feel any substance effect(s), (2) feel high, (3) like the effects, (4) dislike the effects, and (5) want more of the substance by instructing participants to place a mark on a 100mm vertical, visual, analog scale with scores ranging from 0 ="not at all" to 100 = "extremely" for each question. The mean of the individual responses is used to general a total score with a range from 0 to 100, with higher scores indicate a greater "liking" of the effects of the substance. The mean and standard deviation of each treatment condition will be reported.
Time Frame: Study Day 1-3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 45.4 (33.7) | 69.0 (16.7) | 73.2 (14.4)

8. Primary Outcome: Mean Scores on the Marijuana Craving Questionnaire-Short Form (MCQ-SF)
Description: This 12-item multidimensional measure assesses cannabis craving based on 4 factors: Compulsivity, Emotionality, Expectancy, Purposefulness. Each item asks about the respondent's feelings and thoughts about smoking marijuana as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) with higher scores indicating a greater level of craving. The calculation of each subscale is as follows: Compulsivity: Mean of items 2, 7, and 10; Emotionality: Mean of items 4, 6, and 9; Expectancy: Mean of items 5, 11, and 12; Purposefulness: Mean of items 1, 3, and 8 with the minimum possible score = 1 and the maximum possible score = 7 for any subscale. The mean and standard deviation of each subscale for each treatment condition will be reported.
Time Frame: Study Day 1-3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale
  Compulsivity | 2.8 (1.7) | 3.0 (1.8) | 2.5 (1.6)
  Emotionality | 3.1 (2.1) | 3.5 (1.8) | 2.9 (1.9)
  Expectancy | 4.1 (1.8) | 4.6 (1.8) | 3.9 (1.6)
  Purposefulness | 4.6 (1.8) | 4.8 (2.2) | 4.0 (2.3)

9. Primary Outcome: Mean Scores on the Modified Cigarette Evaluation Questionnaire (mCEQ)
Description: The modified Cigarette Evaluation Questionnaire (mCEQ) uses three multi-item subscales and two single items: "Smoking Satisfaction" (items 1, 2, and 12);"Psychological Reward" (items 4 through 8); "Aversion" (items 9 and 10);"Enjoyment of Respiratory Tract Sensations" (item 3); and "Craving Reduction"(item 11). Scores for each subscale are calculated as the mean of the individual item responses or the single item. Higher scores indicate greater intensity on that scale. Items are rated on a seven-point scale ranging from 1 (not at all) to 7 (extremely) and total scores are averaged across all items with a minimum average score of 1 and a maximum average score of 7. Higher scores indicate greater intensity of each smoking effect with, for example, greater satisfaction or psychological reward after smoking. The mean and standard deviation for each treatment condition will be reported.
Time Frame: Study Day 1-3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 1.5 (3.2) | 3.1 (3.5) | 1.4 (1.5)

10. Primary Outcome: Mean Scores on the Positive Affect Negative Affect Schedule (PANAS)
Description: The Positive and Negative Affect Schedule (PANAS) is a brief scale is comprised of 20 items, with 10 items measuring positive affect (e.g., excited, inspired) and 10 items measuring negative affect (e.g., upset, afraid). Each item is rated on a five-point Likert Scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely, to measure the extent to which the affect has been experienced in a specified time frame and the final score is derived out of the sum of the ten items on both the positive and negative side. Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Time Frame: Study Day 1-3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale
  Positive | 26.9 (11.6) | 23.0 (9.6) | 25.8 (11.1)
  Negative | 10.6 (1.2) | 11.4 (3.1) | 10.2 (0.7)

11. Primary Outcome: Mean Scores on the Minnesota Nicotine Withdrawal Scale (MNWS)
Description: The Minnesota Nicotine Withdrawal Scale is an 7-item self - report scale designed to measure the severity of craving and withdrawal symptoms experienced during smoking cessation. Each item is rated on a scale of 0 to 4 with 0=none,1= Slight, 2= Mild, 3= Moderate, and 4=Severe. Seven of the items are symptoms derived from the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) Tobacco Withdrawal diagnosis and are as follows: depression, insomnia, irritability/frustration/anger, anxiety/nervousness, difficulty concentrating, restlessness, increased appetite and at least five of seven items must have responses in order to generate a reliable score. The responses to each item are summed to produce a total withdrawal summary score with greater scores indicating a higher level of severity in nicotine withdrawal symptoms overall. The mean and standard deviation of each treatment condition will be reported with a minimum mean score of 0 and a maximum mean score of 4.
Time Frame: Study Day 1-3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 0.8 (1.0) | 1.2 (1.2) | 0.9 (1.1)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Tobacco Arm | Cannabis Arm | Combined Cannabis and Tobacco Arm
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT02955329/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT02955329/ICF_001.pdf